CLINICAL TRIAL: NCT06427629
Title: Investigator-initiated Exploratory Clinical Trial to Observe Conjunctival Goblet Cell Density Using an Anterior Segment Imaging Device in Patients With Ocular Surface Disease (ODS) and Patients Scheduled for Ocular Surgery Without OSD
Brief Title: Investigator-initiated Clinical Trial to Observe Conjunctival Goblet Cell Using an Anterior Segment Imaging Device
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chang Ho Yoon, Clinical associate professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2311-108-1485
Record Dates: First submitted 2024-05-02; First posted 2024-05-24 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Ocular Surface Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with ocular surface disease (Other): Patients diagnosed with dry eye disease, sjogren syndrome, stevens-johnson syndrome, ocular graft versus host disease.
  Interventions: Device: Imaging of conjunctival goblet cell
- Patients scheduled for ocular surgery without ocular surface disease (Other): Patients without ocular surface disease and scheduled for cataract surgery which requires moxifloxacin administration
  Interventions: Device: Imaging of conjunctival goblet cell

INTERVENTIONS:
Device: Imaging of conjunctival goblet cell — After instillation of moxifloxacin and illuminating with a 405nm light source using confocal fluorescence microscopy, conjunctival goblet cell imaging will be performed in patients with ocular surface disease and patients scheduled for ocular surgery without ocular surface disease

SUMMARY:
Conjunctival goblet cells secrete mucin, vital for tear film stability. Dysfunction can cause tear film issues and lead to diseases like dry eye. Imaging these cells is crucial for diagnosis and treatment. 0.5% moxifloxacin eye drops, an FDA-approved antibiotic, are used to treat bacterial eye infections and prevent infections before surgeries. The investigators developed a non-invasive imaging method for goblet cells, validated in animals, and now plan to test it in humans for diagnosing and treating ocular surface diseases.

DETAILED DESCRIPTION:
Conjunctival goblet cells secrete mucin on the ocular surface, playing a role in forming the mucin layer of the tear film. The mucin layer is crucial for maintaining tear film stability, and dysfunction of conjunctival goblet cells can lead to instability of the mucin layer, causing problems in the tear film. Because various ocular surface diseases stem from tear film instability, imaging of conjunctival goblet cells is essential for diagnosing and treating conditions such as dry eye.

0.5% moxifloxacin eye drops are FDA-approved antibiotics belonging to the quinolone class, widely used to treat bacterial infections in various ocular diseases. Clinically, 0.5% moxifloxacin eye drops are commonly used for purposes such as secondary infection prevention in cases of corneal epithelial defects or perforations caused by ocular surface diseases, as well as for prophylaxis prior to various ophthalmic surgeries, including cataract surgery.

The investigators have previously pioneered non-invasive, high-speed, high-contrast imaging of conjunctival goblet cells. Previous studies have validated the performance and safety of this method by imaging conjunctival goblet cells in mice and rabbit animal models after the instillation of moxifloxacin and illuminating with a 405nm light source using confocal fluorescence microscopy. Furthermore, in this study, the investigators plan to conduct a study involving human subjects to apply our developed conjunctival goblet cell imaging technique for the diagnosis and evaluation of treatment outcomes in ocular surface diseases.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 19 years or older.
* Patients who are currently using or scheduled to use 0.5% moxifloxacin eye drops for ophthalmic surgery (control group) or for ocular surface diseases (patient group: dry eye, Sjogren's syndrome, Stevens-Johnson syndrome, graft versus host disease).
* Patients who have agreed to understand and comply with the clinical trial protocol's plans for medical examinations and follow-up observations.

Exclusion Criteria:

* Pregnant or planning to become pregnant, and lactating women.
* Patients with intellectual disabilities and other psychiatric disorders who, at the discretion of the investigator, are deemed ineligible for participation in the clinical trial.
* Patients with hypersensitivity reactions to 0.5% moxifloxacin eye drops, or patients for whom administration is contraindicated.
* Patients for whom participation in the study is deemed impractical based on the judgment of other medical staff and neutral observers (excluding specified selection/exclusion criteria, based on medical reasons, ethical considerations, low compliance, and understanding of the study).

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Association between conjunctival goblet cell density and severity of dry eye | At the time of imaging
  Severity of dry eye will be assessed based on tear break up time and corneal punctate erosion score

SECONDARY OUTCOMES:
Difference of conjunctival goblet cell density according to disease and additional parameters related with ocular surface disease | At the time of imaging
  Conjunctival punctate erosion score (NEI scale, 0-15), schirmer test (mm), matrix metalloproteinase 9 assay (negative/trace/positive/strong positive), ocular surface disease index (0-100 score) will be assessed as additional parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Chang Ho Yoon, MD PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Changho Yoon, Seoul, South Korea